CLINICAL TRIAL: NCT05822011
Title: Ultrasound Guided Rhomboid Intercostal Subserratus Plane Block Versus Erector Spinae Plane Block in Open Nephrectomy. Randomized Controlled Study
Brief Title: Ultrasound Guided Rhomboid Intercostal Subserratus Plane Block vs Erector Spinae Plane Block in Open Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mahmoud Saad, Assistant Lecturer of Anesthesia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Rhomboid block in nephrectomy
Record Dates: First submitted 2023-03-14; First posted 2023-04-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Post Operative Pain
Keywords: Rhomboid intercostal block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Erector spinae block (Active Comparator): Under strict aseptic precautions, we will begin the scout scan with a high-frequency (6-12 MHz) linear US probe placed parasagitally in cephalocaudal orientation adjacent to C7 spinous process and the first rib will be identified with ultrasound. Then, we can directly count the ribs and come down to desired level of ribs or corresponding transverse process (the 8th thoracic spinous process). Once located, erector spinae and trapezius muscles will be identified overlying it. The skin will be infiltrated by 2 ml of lidocaine 1% subcutaneously and a 22- gauge, 80 mm needle (Stimuplex D, B-Braun, Germany) will be advanced in plane in the cranio-caudal direction. When the needle contacted the transverse process, 1 ml normal saline will be injected to confirm correct needle placement by visualizing the linear pattern of hydrodissection. After aspiration, 30 ml bupivacaine 0.25% will be injected.
  Interventions: Procedure: Erector spinae plane block
- Rhomboid intercostal block (Active Comparator): While the patient in the sitting position, the 5th thoracic spinous process can be identified, a high-frequency (6-12 MHz) linear US probe will be placed in the sagittal plane medial to the medial border of the scapula and then rotated to be 1 to 2 cm medial to the medial scapular border. The plane between the rhomboid major and the intercostal muscles will be identified. 2 ml of lidocaine 1% subcutaneously and a 22- gauge, 80 mm needle (Stimuplex D, B-Braun, Germany) will be advanced in plane from a superomedial to an inferolateral direction then 15 ml of bupivacaine 0.25% will be administered (at the T5 level). Then the probe will be moved caudally and laterally to identify the tissue plane between the serratus anterior and the external intercostal muscle at the T8 level. The needle will be directed caudally and laterally beyond the inferior angle of the scapula. 15 ml of bupivacaine 0.25% will be administered.
  Interventions: Procedure: Rhomboid intercostal subserratus plane block

INTERVENTIONS:
Procedure: Rhomboid intercostal subserratus plane block — Fascial plane block
  Other Names: RISS
  Arms: Rhomboid intercostal block
Procedure: Erector spinae plane block — Fascial plane block
  Other Names: ESB
  Arms: Erector spinae block

SUMMARY:
Our aim is to measure the efficacy of rhomboid intercostal subserratus plane block and erector spinae plane block in patients undergoing open nephrectomy

DETAILED DESCRIPTION:
Open nephrectomy incision is associated with a high incidence of intense immediate postoperative pain and chronic pain the months following surgery. Regional anesthesia techniques are commonly recommended for pain management in open nephrectomy as they decrease parenteral opioid requirements and improve patient satisfaction. Rhomboid intercostal subserratus plane block (RISS) is considered a novel approach for chest wall and upper abdominal analgesia, initially showed promising results, first reported in 2016. Erector Spinae Plane block (ESB), was initially described in 2016 for analgesia in thoracic neuropathic pain. It has also been widely used in both adults and children at different levels for different indications. Epidural analgesia is the gold standard for perioperative analgesia in open surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Type of surgery; open nephrectomy.
2. Physical status ASA II, III.
3. Body mass index (BMI): > 20 kg/ m2 and < 35 kg/ m2.

Exclusion Criteria:

1. Patient refusal.
2. Local infection at the puncture site.
3. Severe respiratory or cardiac disorders.
4. Advanced liver or kidney disease.
5. History of psychological disorders and/or chronic pain.
6. Contraindication to regional anesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
7. Patients with known sensitivity or contraindication to amide local anesthetics used in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine consumption in (mg) | first 24 hours postoperatively.
  amount of morphine in mg consumed in 1st 24 hours

SECONDARY OUTCOMES:
Time of first request of analgesia | first 24 hours postoperatively
  calculated from the time of complete injection of local anesthetics till the numerical pain rating scale (NRS) is ≥3.(NRS requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable)
Total amount fentanyl in (microgram) | intra operative duration
  total amount of intraoperative fentanyl consumed in micrograms
Change in heart rate in (beat/min) | From just before induction till 24 hours post operatively
  Readings will be taken as baseline preoperative reading, immediately after surgical incision and at 15-minute intervals intraoperatively and 30 minutes,2,4,8,12,16 and 24 hours postoperatively
Change in mean arterial blood pressure in (mmHg) | From just before induction till 24 hours post operatively
  Readings will be taken as baseline preoperative reading, immediately after surgical incision and at 15-minute intervals intraoperatively and 30 minutes,2,4,8,12,16 and 24 hours postoperatively
Numeric Pain Rating Scale | first 24 hours postoperatively
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable
Nausea and vomiting Scores | first 24 hours postoperatively
  Nausea and vomiting Scores using a four-point verbal scale. (None =no nausea, mild =nausea but no vomiting, moderate=vomiting one attack, severe =vomiting >one

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Al Awad, Professor, Study Chair — National Cancer Institute (NCI)
Locations (1):
- National Cancer Institute, Cairo, Egypt

REFERENCES:
- [Background] Bravi CA, Larcher A, Capitanio U, Mari A, Antonelli A, Artibani W, Barale M, Bertini R, Bove P, Brunocilla E, Da Pozzo L, Di Maida F, Fiori C, Gontero P, Li Marzi V, Longo N, Mirone V, Montanari E, Porpiglia F, Schiavina R, Schips L, Simeone C, Siracusano S, Terrone C, Trombetta C, Volpe A, Montorsi F, Ficarra V, Carini M, Minervini A. Perioperative Outcomes of Open, Laparoscopic, and Robotic Partial Nephrectomy: A Prospective Multicenter Observational Study (The RECORd 2 Project). Eur Urol Focus. 2021 Mar;7(2):390-396. doi: 10.1016/j.euf.2019.10.013. Epub 2019 Nov 12. PMID 31727523
- [Background] Saleh AH, Abdallah MW, Mahrous AM, Ali NA. Quadratus lumborum block (transmuscular approach) versus transversus abdominis plane block (unilateral subcostal approach) for perioperative analgesia in patients undergoing open nephrectomy: a randomized, double-blinded, controlled trial. Braz J Anesthesiol. 2021 Jul-Aug;71(4):367-375. doi: 10.1016/j.bjane.2021.01.009. Epub 2021 Mar 21. PMID 33762197
- [Background] Kang XH, Bao FP, Xiong XX, Li M, Jin TT, Shao J, Zhu SM. Major complications of epidural anesthesia: a prospective study of 5083 cases at a single hospital. Acta Anaesthesiol Scand. 2014 Aug;58(7):858-66. doi: 10.1111/aas.12360. Epub 2014 Jun 24. PMID 24961586
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] Chin KJ, Adhikary S, Sarwani N, Forero M. The analgesic efficacy of pre-operative bilateral erector spinae plane (ESP) blocks in patients having ventral hernia repair. Anaesthesia. 2017 Apr;72(4):452-460. doi: 10.1111/anae.13814. Epub 2017 Feb 11. PMID 28188621
- [Background] Ueshima H, Otake H. RETRACTED: Erector spinae plane block provides effective pain management during pneumothorax surgery. J Clin Anesth. 2017 Aug;40:74. doi: 10.1016/j.jclinane.2017.04.016. Epub 2017 Apr 28. No abstract available. PMID 28625453
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292
- [Background] Oh SK, Lim BG, Won YJ, Lee DK, Kim SS. Analgesic efficacy of erector spinae plane block in lumbar spine surgery: A systematic review and meta-analysis. J Clin Anesth. 2022 Jun;78:110647. doi: 10.1016/j.jclinane.2022.110647. Epub 2022 Jan 11. PMID 35030493
- [Background] Elsharkawy H, Maniker R, Bolash R, Kalasbail P, Drake RL, Elkassabany N. Rhomboid Intercostal and Subserratus Plane Block: A Cadaveric and Clinical Evaluation. Reg Anesth Pain Med. 2018 Oct;43(7):745-751. doi: 10.1097/AAP.0000000000000824. PMID 30169476
- [Background] Elsharkawy H, Saifullah T, Kolli S, Drake R. Rhomboid intercostal block. Anaesthesia. 2016 Jul;71(7):856-7. doi: 10.1111/anae.13498. No abstract available. PMID 27291611
- [Background] Elsharkawy H, Pawa A, Mariano ER. Reply to Dr Price: Interfascial plane blocks - a Time to Pause. Reg Anesth Pain Med. 2019 Jan;44(1):138. doi: 10.1136/rapm-2018-100020. Epub 2018 Dec 19. No abstract available. PMID 30640671
- [Background] Sharma SK, Mistry T, Ahmed S. Ultrasound-guided thoracic erector spinae plane block: A modified transverse approach. Saudi J Anaesth. 2020 Jan-Mar;14(1):142-143. doi: 10.4103/sja.SJA_624_19. Epub 2020 Jan 6. No abstract available. PMID 31998046
- [Background] Elsharkawy H, Hamadnalla H, Altinpulluk EY, Gabriel RA. Rhomboid intercostal and subserratus plane block -a case series. Korean J Anesthesiol. 2020 Dec;73(6):550-556. doi: 10.4097/kja.19479. Epub 2020 Feb 12. PMID 32046475
- [Background] Lichtenstein D, van Hooland S, Elbers P, Malbrain ML. Ten good reasons to practice ultrasound in critical care. Anaesthesiol Intensive Ther. 2014 Nov-Dec;46(5):323-35. doi: 10.5603/AIT.2014.0056. PMID 25432552
- [Background] Apfel CC, Kranke P, Eberhart LH, Roos A, Roewer N. Comparison of predictive models for postoperative nausea and vomiting. Br J Anaesth. 2002 Feb;88(2):234-40. doi: 10.1093/bja/88.2.234. PMID 11883387
- [Background] Sakae TM, Yamauchi LHI, Takaschima AKK, Brandao JC, Benedetti RH. [Comparison between erector spinal plane block and epidural block techniques for postoperative analgesia in open cholecystectomies: a randomized clinical trial]. Braz J Anesthesiol. 2020 Jan-Feb;70(1):22-27. doi: 10.1016/j.bjan.2019.12.009. Epub 2020 Feb 27. PMID 32171499
- [Derived] Eltwab DA, Abed SM, Saad A, Aliem MAA, Elsamahy KA, Elshamy FH, Gad AF, Elsabeeny WY. Ultrasound-guided erector spinae plane block versus rhomboid intercostal sub-serratus plane block for postoperative analgesia in open radical nephrectomy: a randomized clinical study. BMC Anesthesiol. 2025 Oct 22;25(1):514. doi: 10.1186/s12871-025-03377-4. PMID 41120933